CLINICAL TRIAL: NCT03888196
Title: Evaluation of the Efficacy of Panax Ginseng on Lipid Metabolism in Men and the Relationship With Sports Practice.
Acronym: GinsengRun
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, José Serrano, Principal Investigator, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nutren-Disanta 0012018
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Sports Physical Therapy
Keywords: Panax; Lipid Metabolism; Sport Performance; Running; Ginseng

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 500 mg/day of Panax Ginseng. 2 weeks treatment
  Interventions: Dietary Supplement: Panax Ginseng Supplementation
- Control Group (Placebo Comparator): 500 mg/day of Celulose. 2 weeks treatment
  Interventions: Dietary Supplement: Placebo Supplementation

INTERVENTIONS:
Dietary Supplement: Panax Ginseng Supplementation — 500 mg/day of Panax Ginseng
  Arms: Intervention Group
Dietary Supplement: Placebo Supplementation — 500 mg/day of Cellulose
  Arms: Control Group

SUMMARY:
Panax Ginseng (P ginseng), C.A. Meyer, Red, Chinese or Korean ginseng is a plant from eastern Asia and is one of the most widely used herbal products in the world. P ginseng has been been used for many years for different medical therapies. Previous studies have demonstrate that P. ginseng root extract supplementation may promote fat oxidation, increase hepatic glycogen levels and produce a glycogen-sparing and antifatigue effect during exercise in swimming rats. Notwithstanding, although there is some evidence of P. ginseng effects in humans, no evidence has been obtained respect to its supplementation in human sport performance. The aim of this study is to assess the effect of P ginseng extract supplementation on the lipid metabolism and sport performance in male endurance runners. For this purpose, the effect of supplementation for 2 weeks of 500 mg/day of P. ginseng will be evaluated in a sub-maximal physical stress test. Variables of lipid metabolism, energy consumption, fatigue, and endurance will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Athletic men of aerobic type, who participate in a supervised training as a previous step to the accomplishment of competitions
* Which their age is older than 18 years
* Training superior or equal to 3 days per week and that these workouts are stable during the intervention.

Exclusion Criteria:

* Athletes with high blood pressure, with pharmacological treatment for hypercholesterolemia, diabetes, any psychiatric illness
* Athletes who practice sports without having the objective of increasing sports performance
* Athletes who use some type of ergogenic sport supplementation looking to optimize any aspect related to the sport.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline plasmatic Total Lipids at 2 weeks | 2 weeks
  Total Lipids in the plasma are measured in mg / dL
Change from baseline plasmatic Triglycerides at 2 weeks | 2 weeks
  Triglycerides in the plasma are measured in mg / dL
Change from baseline Respiratory Exchange Rate at 2 weeks | 2 weeks
  To quantify the amount of Oxygen consumed and the amount of carbon dioxide produced. (mL/Kg/Min)

CONTACTS AND LOCATIONS:
Overall Officials: Jose D Serrano, Dr, Study Chair — Universitat de Lleida; Alba Naudí, Dra, Study Director — Universitat de Lleida; Cristian D Hernandez, PhD Student, Principal Investigator — Universitat de Lleida

IPD SHARING:
Plan to Share IPD: No